CLINICAL TRIAL: NCT04288128
Title: Integrated Functional Evaluation of the Cerebellum
Acronym: CERMOI
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Biogen (Industry); Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C18-29; 2018-A02563-52 (Registry Identifier: Secondary ID)
Record Dates: First submitted 2020-02-17; First posted 2020-02-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-01

CONDITIONS: Spinocerebellar Ataxia Type 2; Spinocerebellar Ataxia Type 7
Keywords: Spinocerebellar ataxia; Multimodal approach; Biomarker; Antisense oligonucleotides (ASOs) therapy
MeSH Terms: conditions — Spinocerebellar Ataxias | interventions — Spinal Puncture; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood collected for DNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SCA early-manifest and premanifest patients: This cohort is defined by individuals with a SARA score between 0 and 15 (both values included).
  Interventions: Procedure: Lumbar puncture; Other: Magnetic Resonance Imaging (MRI)
- Control participants: This cohort is defined by individuals with a SARA score less than 5 and no significant neurological symptoms.
  Interventions: Procedure: Lumbar puncture; Other: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: Lumbar puncture — Each participant will undergo lumbar puncture at first visit (M0) and last visit (M12)
Other: Magnetic Resonance Imaging (MRI) — Each participant will undergo scanning at 3 visits (M0, M6 and M12)

SUMMARY:
One of the main objectives of this project is to validate potential biological, clinical and/or imaging biomarkers in SCA patients through a multimodal assessment, for future ASOs trials.

DETAILED DESCRIPTION:
Spinocerebellar ataxias (SCAs) are autosomal dominantly inherited neurological disorders, characterized by a predominant atrophy of the cerebellum and the brainstem. The most common forms are caused by abnormal CAG repeat expansions, encoding elongated polyglutamine (polyQ).

Nowadays, no preventive or curative treatments are available but different therapeutic approaches are ongoing. Antisense oligonucleotides (ASOs) therapy showed promising results in Huntington disease (HD), a disease that shares with the SCAs the same mutational mechanism. ASOs are currently under development for SCAs.

However, in SCAs, clinical scales as an only criteria to monitor a treatment are not appropriate because of the lack of sensitivity of change and the small number of patients available. The importance to dispose of outcome measures to inform about the efficacy of a treatment is fundamental as well as of new alternative designs to conduct a clinical trial in rare diseases with small sample sizes.

A comprehensive, multimodal approach is hence needed to provide a translational and integrated overview of cerebellar dysfunction in polyQ SCAs over a year.

ELIGIBILITY:
Common inclusion criteria for all participants:

* Ability to walk independently 30 foot without an assistive device
* Able to stand unassisted for 30 seconds
* Affiliated with the French social security, or a social security equivalent, if they are not French.
* Capacity to consent
* Signed Informed Consent by the subject
* Ability to undergo MRI scanning

Inclusion criteria for SCA patients:

* Genetic diagnosis of SCA 2 or 7 (available CAG repeat length)
* SARA score ≤15

Inclusion criteria for control participants:

* Negative Genetic diagnosis of SCA2/SCA7 available
* No significant neurological symptoms
* SARA score < 5

Common inclusion criteria for elective participant for CSF sampling:

• Ability to undergo a lumbar puncture

Exclusion criteria

* Subjects currently receiving, or having received within 2 months prior to enrolment into this study, any investigational drug
* Pregnancy or breastfeeding
* Genotype consistent with other inherited ataxias
* Changes in coordinative physical and occupational therapy for ataxia 2 months prior to study participation
* Concomitant disorder(s) or condition(s) that affects assessment of ataxia or severity of ataxia during this study
* Contra-indications to MRI examination
* Person deprived of their liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Early stage subjects and premanifest mutation carriers refer to individuals who tested positive for the SCA 2 or 7 gene mutation and SARA score between 0 and 15 (both values included)
  2. Control participants refer to individuals with non-mutation carriers.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Identification of biological, clinical and/or imaging biomarkers in SCA2 and SCA7 patients mutations carriers and patients through a multimodal assessment over one year to prepare therapeutic trials | Over one year

SECONDARY OUTCOMES:
To determine the cross-sectional and longitudinal variability of SARA (Scale for the Assessment and Rating of Ataxia) and CCFS (Composite Cerebellar Functional Score) scores in SCA 2 and SCA 7 gene mutation carriers and healthy controls over one | Over one year
Determine the cross-sectional and longitudinal variability of volumetric MRI and NMR-proto spectroscopy in SCA 2 and SCA 7 gene mutation carriers and healthy controls | Over one year
Delineate a specific pattern of frontal-like cognitive deficit in SCAs gene carriers | Over one year
  Evolution of neuropsychological scores and Cerebellar Cognitive Affective/Schmahmann Syndrome Scale. The neuropsychological data collected has to evaluate the cerebellar cognitive affective syndrome (CCAS). The CCAS consisting of cognitive and affective deficits due to cerebellar disease.
To determine the cross-sectional and longitudinal variability of CSF, blood and urine biomarkers in SCAs gene mutation carriers and controls | Over one year
  eg. specific mutant protein dosage in CSF sample for each genotype over 1 year, if available
To explore the relationship of CSF, blood and urine biomarker levels in relation to clinical and imaging markers of disease progression | Over one year
To assess the feedback of individuals for the disease (Most bothersome symptoms) | Over one year
  Evolution of a Most Bothersome Symptom (MBS) questionnaire will be performed by the physician in order to determine patients' most bothersome symptoms. This qualitative report investigating the subjective complaint and feedback of patients
To assess the feedback of individuals for the disease thanks to quality of life questionnaires | Over one year
  Evolution of quality of life self-administrated questionnaires :
  Patient global impression: is a global index that may be used to rate the response of a condition EQ-5D is a standardized instrument which measures health-related quality of life that can be used in a wide range of health conditions and treatments Patient Health Questionnaire (PHQ 9) is a self-administered depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
To determine the cross-sectional and longitudinal variability of quantitative measures of postural stability, free walking and turning in SCA 2 and SCA 7 mutation carriers and healthy controls | Over one year
  Evolution of postural sway measures from the sternum and the lumbar spine by wearable APDM® sensors and evolution of cerebellar instability by Fitbit® smartwatch
To determine the cross-sectional and longitudinal variability of quantitative measures of oculomotor recording in SCA 2 and SCA 7 gene mutations carriers and healthy controls. | Over one year
To determine the cross-sectional and longitudinal variability of optical coherence tomography in SCA 2 and SCA 7 gene mutations carriers | Over one year
To determine the cross-sectional and longitudinal variability of adaptative optics in SCA 2 and SCA 7 gene mutations carriers | Over one year
To determine the cross-sectional and longitudinal variability of autofluorescence, visual acuity, in SCA 2 and SCA 7 gene mutations carriers | Over one year
To determine the cross-sectional and longitudinal variability of visual field in SCA 2 and SCA 7 gene mutations carriers | Over one year
To determine the cross-sectional and longitudinal variability of colour contrast sensitivity in SCA 2 and SCA 7 gene mutations carriers | Over one year
To determine the cross-sectional and longitudinal variability of electroretinogram in SCA 2 and SCA 7 gene mutations carriers | Over one year
To determine the cross-sectional and longitudinal variability of static perimetry in SCA 2 and SCA 7 gene mutations carriers | Over one year
To determine the cross-sectional and longitudinal variability of visual evoked potential in SCA 2 and SCA 7 gene mutations carriers | Over one year

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra DURR, Principal Investigator — Institut du Cerveau - Paris Brain Institute
Locations (1):
- Institut du Cerveau - Paris Brain Institute, Paris, France

REFERENCES:
- [Result] Coarelli G, Dubec-Fleury C, Petit E, Sayah S, Fischer C, Nassisi M, Gatignol P, Dorgham K, Daghsen L, Daye P, Cunha P, Kacher R, Hilab R, Hurmic H, Lamaziere A, Lamy JC, Welter ML, Chupin M, Mangin JF, Lane R, Gaymard B, Pouget P, Audo I, Brice A, Tezenas du Montcel S, Durr A. Longitudinal Changes of Clinical, Imaging, and Fluid Biomarkers in Preataxic and Early Ataxic Spinocerebellar Ataxia Type 2 and 7 Carriers. Neurology. 2024 Sep 10;103(5):e209749. doi: 10.1212/WNL.0000000000209749. Epub 2024 Aug 12. PMID 39133883
- [Result] Nassisi M, Coarelli G, Blanchard B, Dubec-Fleury C, Drine K, Kitic N, Sancho S, Hilab R, Tezenas du Montcel S, Junge C, Lane R, Arnold HM, Durr A, Audo I. ATXN7-Related Cone-Rod Dystrophy: The Integrated Functional Evaluation of the Cerebellum (CERMOI) Study. JAMA Ophthalmol. 2024 Apr 1;142(4):301-308. doi: 10.1001/jamaophthalmol.2024.0001. PMID 38421662